CLINICAL TRIAL: NCT06065657
Title: Effect of Nutritional Ketosis on Alcohol Metabolism
Acronym: KAM
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 853707; 24446 (Other Grant/Funding Number: UPenn ITMAT); R21AA031088-01A1 (NIH)
Record Dates: First submitted 2023-09-20; First posted 2023-10-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ketoses, Metabolic; Ketogenic Dieting; Alcohol Intoxication; Magnetic Resonance Imaging; Alcohol Drinking
Keywords: Ketone supplement
MeSH Terms: conditions — Ketosis; Alcoholic Intoxication; Alcohol Drinking | interventions — Diet, Ketogenic; Ethanol

STUDY DESIGN:
Intervention Model Description: Three-way, open-labeled, crossover trial in which participants will undergo three alcohol tolerance tests, each following a 3-days dietary intervention: (1) control diet (~ 50% kcal carbohydrates), (2) ketogenic diet (~5-10% kcal carbohydrates), and (3) control diet with 3x daily administration of 10 g Ketone Supplement (KS) drink (30 g/day, Kenetik: ketone Drink, VitaNav Inc., Washington D.C.).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ketogenic diet (Experimental): Eat a ketogenic diet for 3 days
  Interventions: Drug: Ethanol
- Control Diet (Placebo Comparator): Eat a control diet for 3 days
  Interventions: Drug: Ethanol
- Ketone supplement (Experimental): Eat a control diet for 3 days with a ketone supplement drink
  Interventions: Other: Control Diet; Drug: Ethanol
- Alcohol Intervention (Experimental): Alcohol lab, participants will receive ethanol drinks that are dose-adjusted for body weight and sex differences in pharmacokinetics and calculated to obtain a final breath alcohol concentration of 0.08%
  Interventions: Dietary Supplement: Ketone Supplement; Other: Control Diet; Other: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketone Supplement — Ketone supplement 3x day with control diet for 3 days.
  Other Names: D-Beta-hydroxybutyric acid and R-1,3 butanediol
  Arms: Alcohol Intervention
Other: Control Diet — Control Diet breakfast, lunch, and dinner for 3 days.
  Other Names: ~ 50% kcal carbohydrates diet
  Arms: Alcohol Intervention; Ketone supplement
Other: Ketogenic diet — Ketogenic Diet breakfast, lunch, and dinner for 3 days.
  Other Names: ~5-10% kcal carbohydrates diet
  Arms: Alcohol Intervention
Drug: Ethanol — After 3 days of diet intervention, participants will receive alcohol drinks that dose-adjusts for body weight and sex differences in pharmacokinetics and calculated to obtain a final breath alcohol concentration of 0.08%
  Other Names: Alcohol
  Arms: Control Diet; Ketogenic diet; Ketone supplement

SUMMARY:
The research study is being conducted in health controls to better understand the effects of ketosis on brain functioning after 3 different, randomly assigned, 3-day dietary interventions and the acute effects of alcohol after consuming about 4-5 alcohol beverages. The labs visits will use magnetic resonance imaging (MRI) scans to study the brain, measuring levels of nicotinamide adenine dinucleotide (NAD), lactate, neurotransmitters glutamate, and Gamma-aminobutyric acid (GABA).

DETAILED DESCRIPTION:
The research study is being conducted to better understand the effects of ketosis on brain functioning and the acute effects of alcohol. Healthy participants will undergo three randomly assigned dietary interventions, each lasting three days, followed by a study lab visit day on day 4. The three interventions are: (1) Eat a ketogenic diet for 3 days, (2) eat a control diet for 3 days with a ketone supplement drink, and (3) eat a control diet for 3 days. The dietary interventions will be spaced 1 week apart. The ketone supplement drink "bis-octanoyl (R)-1,3-butanediol" (Kenetik: Ketone Drink, VitaNav Inc., Washington D.C.) 12.5g of ketones, TID PO (by mouth).) is a dietary supplement that has been extensively studied in humans and is designated by the FDA as Generally Recognized as Safe (GRAS). Its use in this study is experimental. On the day of the 3 labs visits days, magnetic resonance imaging (MRI) will be used to study the brain. Specifically, levels of nicotinamide adenine dinucleotide (NAD) (a coenzyme that is important for energy metabolism), lactate (a metabolite produced during energy metabolism), and neurotransmitters glutamate and GABA. Following the scans, participants will be provided a dose of alcohol that will elevate participants breath alcohol levels to approximately 0.08% to measure the acute effects of alcohol.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide signed, informed consent and commit to completing study procedures.
2. Reported on at least one day in the month prior to consent of consuming 2 or more standard alcohol drinks on a single day.

Exclusion Criteria:

1. Unwilling or unable to refrain from use, within 24 hours of the alcohol lab procedures, psychoactive medications or medication that may affect study results.
2. Current Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of any major psychiatric disorder (other than nicotine use disorders, or marijuana use disorders) as identified by clinical examination or structured interview that could interfere with study participation or make it hazardous for the subject.
3. Currently taking medication(s) that could interfere with study participation or make it hazardous for the subject to participate. (e.g. anticholinergics; antipsychotics; lithium; psychotropic drugs not otherwise specified)
4. Positive urine drug screen, positive for all substances but marijuana at screening or study visits (may be repeated once and if the result is negative on repeat, it is not exclusionary).
5. A current, clinically significant physical disease or abnormality on the basis of medical history, or routine laboratory evaluation that can impact brain function, the use of a ketone supplement, administration of ketogenic diet, or the use of alcohol (e.g., epilepsy, diabetes, irritable bowel syndrome, Crohn's disease, liver disease, kidney disease, kidney stones, chronic metabolic acidosis or a cardiomyopathy as determined by history and clinical exam).
6. Currently suffering from or has a history of stroke and/or stroke related spasticity.
7. Head trauma with loss of consciousness for more than 30 minutes or associated with skull fracture, inter-cranial bleeding or abnormal MRI (self-report, medical history).
8. Weight greater than 225lbs (Need to cap amount of alcohol given based on weight to individuals).
9. Females who are pregnant or breast-feeding
10. Contraindication to MRI, including presence of ferromagnetic objects, claustrophobia or fear of enclosed, medical conditions that prevent subjects from lying comfortably flat on his/ her back for up to 2 hrs.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in breath alcohol concentration | 3 hours
  Breath alcohol concentration measured in mg/L of air. The range is .000 to .400 g/L. Change in breath alcohol concentration, pre to post alcohol consumption after 3 day diet intervention during lab day.

SECONDARY OUTCOMES:
Change in motor agility tasks | 3 hours
  Motor agility will be assessed with the grooved pegboard task, in which participants will place pegs onto a metal surface containing 25 keyhole-shaped holes that differ in orientation. Measured in seconds, range 0 to 5 minutes. Change in motor agility tasks pre to post alcohol consumption after 3 day diet intervention.
Change in cognitive performance tasks | 3 hours
  Cognitive performance will be measured with a cued go/no-go task, in which participants will press a computer keyboard key in response to a "go" target and suppress the action in response to a "no-go" target. Measured in % correct responses 0-100. Pre to post alcohol consumption after 3 day diet intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Corinde Wiers, Ph.D., Principal Investigator — University of Pennsylvania; Henry Kranzler, MD, Study Director — University of Pennsylvania; Kyle Kampman, MD, Study Director — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania, United States